CLINICAL TRIAL: NCT06043310
Title: Effects of Continuous Estrogen on Human in Vivo Microvascular Function
Brief Title: Estrogen and Microvascular Function
Status: Active, not recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Julie K. Freed, Associate Professor, Medical College of Wisconsin
Other Study IDs: PRO40920
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Estrogen; Cardiovascular Diseases; Microvasculature; Oral Contraceptive Use
Keywords: Female; oral contraceptive
MeSH Terms: conditions — Cardiovascular Diseases | interventions — NG-Nitroarginine Methyl Ester; Acetylcholine; Nitroprusside

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Continuous estrogen/progestin: Females who have had continuous estrogen/progestin treatment for a minimum of 1 year.
  Interventions: Drug: Nω-nitro-L-arginine methyl ester (L-NAME); Drug: Acetylcholine; Drug: Sodium Nitroprusside
- No Estrogen/progestin: Females who have not had continuous estrogen treatment for a minimum of 5 years.
  Interventions: Drug: Nω-nitro-L-arginine methyl ester (L-NAME); Drug: Acetylcholine; Drug: Sodium Nitroprusside
- Continuous progestin: Females who have had continuous progestin treatment for a minimum of 1 year.
  Interventions: Drug: Nω-nitro-L-arginine methyl ester (L-NAME); Drug: Acetylcholine; Drug: Sodium Nitroprusside

INTERVENTIONS:
Drug: Nω-nitro-L-arginine methyl ester (L-NAME) — L-NAME will be infused locally through microdialysis catheters.
Drug: Acetylcholine — ACh will be infused locally through microdialysis catheters.
Drug: Sodium Nitroprusside — SNP will be infused locally through microdialysis catheters.

SUMMARY:
The goal of this study is to learn how long-term use of estrogen affects blood vessels in healthy adults.

Participants will:

* give one blood draw of 5 mL
* have one Dexa Scan taken to measure adipose and muscle mass
* have a camera placed under the tongue to take pictures of blood vessels
* have 2 laser Doppler microdialysis catheters placed on the forearm to monitor blood vessels before and after local drug infusion

Researchers will compare blood vessel function of those who take estrogen to those who do not.

ELIGIBILITY:
Inclusion Criteria:

Estrogen/Progestin Group

* Adults aged 18-40 years
* Females with estrogen/progestin treatment for a minimum of 1 year.
* Blood pressure <140/ < 90 mmHg
* No more than 1 cardiovascular risk factor Control Groups
* Adults aged 18-40 years
* Female with no estrogen/progestin treatment for minimum of 5 years.
* Female undergoing progestin only treatment for a minimum of 1 year.
* Blood pressure <140/ < 90 mmHg
* No more than 1 cardiovascular risk factor

Exclusion Criteria:

* Medications that could alter cardiovascular control
* Rash, skin disease, or pigmentation disorders on both forearms
* Anemia
* Kidney Disease
* Known skin allergies
* Smoking or tobacco use within last 6 months
* Coronary Artery Disease

  -1 cardiovascular risk factor Hypertension Diabetes Hypercholesterolemia Hyperlipidemia
* Bleeding disorders
* Use of anti-coagulants
* Allergies to study drugs
* Use of topical/non-topical steroids in last 6 months
* Internal mouth sores
* Forearms covered with tattoos
* Pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Change in blood vessel dilation | 2 hours
  Cutaneous vascular conductance in response to acetylcholine, L-NAME, and sodium nitroprusside infusions will be calculated as percentage of cardiovascular conductance.
Change in Perfused Vessel Density | 0.5 hours
  Total vessel density (TVD) will be calculated using the DeBacker Score manual analysis on all images that have a minimum microcirculation image quality score (MIQS) of 10. Perfused vessel density (PVD) will be calculated by multiplying total vessel density (TVD) x proportion of perfused vessels (PPV%).

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Wauwatosa, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided